CLINICAL TRIAL: NCT04983472
Title: Comparison of Respiratory Muscle Activations During Dyspnea Reduction Positions in Individuals With Chronic Obstructive Pulmonary Disease
Brief Title: Comparison of Respiratory Muscle Activations During Dyspnea Reduction Positions in Individuals
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ceyhun Topcuoğlu, Research Assistant, Abant Izzet Baysal University
Other Study IDs: AIBU-FTR-CT-01
Record Dates: First submitted 2021-07-09; First posted 2021-07-30 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; Surface Electromyography; Ventilation; Dyspnea
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Aspiration; Dyspnea | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational Group: Individuals diagnosed with Chronic Obstructive Pulmonary Disease by the Department of Pulmonology of the Faculty of Medicine of Bolu Abant Izzet Baysal University will be referred to the Department of Physiotherapy and rehabilitation of the Faculty of Health Sciences of Bolu Abant Izzet Baysal University
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Respiratory muscle electromyographic activations of individuals will be taken during supine, normal sitting and dyspnea reduction positions. Individuals with chronic obstructive pulmonary disease will be asked to perform normal breathing, pursed lip breathing, and breathing control during these positions. Respiratory muscle activation measurement of individuals will be taken during different breathing patterns in each position. Respiratory functions will be evaluated with pulmonary function test, respiratory muscle strength, intraoral pressure measurement device, respiratory muscle activation with surface electromyographic device, health status disorder with Chronic Obstructive Pulmonary Disease Assessment Scale, dyspnea with Modified Medical Research Council Dyspnea Scale and Modified Borg Scale. Participants' names, anthropometric measurements, demographic data, contact information and medical history will be collected and recorded with the patient anamnesis form.

SUMMARY:
Chronic and progressive dyspnea is the most characteristic symptom of chronic obstructive pulmonary disease. There are studies in the literature showing that electromyography activations of respiratory muscles increase in individuals with chronic obstructive pulmonary disease and that the severity of the perceived shortness of breath is associated with muscle activation. However, no study has been found comparing respiratory muscle activations during pursed lip breathing and normal breathing in the dyspnea reduction positions and supine position used in the treatment and management of chronic obstructive pulmonary disease. The aim of this study is to evaluate the effects of different dyspnea reduction positions on respiratory muscle activations separately, to compare respiratory muscle activation during normal breathing, respiratory control and pursed lip breathing during these different positions, and to classify muscle activations according to the severity of chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease is a common, preventable and treatable disease characterized by persistent respiratory symptoms and airway limitation due to airway and/or alveolar abnormality, which is affected by many factors that cause abnormal lung development resulting from exposure to harmful gases or particles. Chronic obstructive pulmonary disease is known as the fourth most common cause of death in the world and is expected to rise to third place by the end of 2020. Physiopathological changes such as airflow limitation, bronchial fibrosis, increased airway resistance, ciliary dysfunction, gas exchange abnormalities and air trapping occur in chronic obstructive pulmonary disease. While smoking is the most common risk factor in chronic obstructive pulmonary disease; Occupational dust and chemicals, air pollution, lung growth and development, genetic predisposition such as age and gender, and exposure to environmental effects. Symptoms such as shortness of breath (dyspnea), cough, and sputum are common in chronic obstructive pulmonary disease.

Chronic and progressive dyspnea is the most characteristic symptom of chronic obstructive pulmonary disease. About 30% of individuals with chronic obstructive pulmonary disease have a productive cough. These symptoms can vary from day to day and may precede airflow limitation for years. Significant airflow limitation may also be present without chronic dyspnea, cough, and sputum production. Although chronic obstructive pulmonary disease is defined based on air restriction, individuals with chronic obstructive pulmonary disease usually make the decision to seek treatment based on the effect of symptoms on functional status. Dyspnea, which is the main symptom of chronic obstructive pulmonary disease, is the main cause of disability and anxiety associated with the disease. Typical chronic obstructive pulmonary disease patients define dyspnea as a feeling of increased breathing effort, heaviness in the chest, and air hunger.

Today, it has been shown that there are many underlying causes of dyspnea. In chronic obstructive pulmonary disease patients, minute ventilation and dead space ventilation due to increased workload increase respiratory motor output in association with an increase in carbon dioxide production. As a result, individuals feel short of breath. Simple mechanical distention of the airways during exhalation, which is defined as dynamic airway compression, is another cause of dyspnea in patients with chronic obstructive pulmonary disease. Different positions and breathing patterns affect the perception of dyspnea in individuals with chronic obstructive pulmonary disease. In current studies, individuals with chronic obstructive pulmonary disease have an increased perception of shortness of breath in the supine position (orthopnea); It was observed that the perception of shortness of breath decreased in pursed lib (pursed lip) breathing and dyspnea reduction positions. Therefore, pursed lip breathing and breathlessness reduction positions are frequently used in the treatment of individuals with chronic obstructive pulmonary disease. Leaning forward, comfortable sitting, leaning forward, standing with the back leaning, high side lying are the most commonly used positions to reduce dyspnea.

It has been shown that the forward bending position, one of the dyspnea-reducing positions, improves the length-tension relationship and function of the diaphragm muscle, decreases the activity of the sternocleidomastoideus, scalene muscles, improves thoracoabdominal movement, and helps to reduce shortness of breath. Pursed-lip breathing, on the other hand, increases tidal volume, leading to increased rib cage movement and accessory muscle recruitment during inspiration and expiration.

Compared to healthy individuals, individuals with chronic obstructive pulmonary disease have an increased electromyographic activation of respiratory muscles. In chronic obstructive pulmonary disease patients, there is an increase in respiratory muscle activation and shortness of breath due to the imbalance between the workload and capacity of the respiratory muscles. In current studies, it has been observed that the severity of dyspnea perception and respiratory muscle activations are related.

There are studies in the literature showing that electromyographic activations of respiratory muscles increase in individuals with chronic obstructive pulmonary disease and that the severity of the perceived shortness of breath is associated with muscle activation. However, no study has been found comparing respiratory muscle activations during pursed lip breathing and normal breathing in dyspnea reduction positions and supine position used in the treatment and management of chronic obstructive pulmonary disease. The aim of this study is to evaluate the effects of different dyspnea reduction positions on respiratory muscle activations separately, to compare respiratory muscle activation during normal breathing, respiratory control and pursed lip breathing during these different positions, and to classify muscle activations according to the severity of chronic obstructive pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with chronic obstructive pulmonary disease
* Be between the ages of 40-65
* No medication changes due to acute exacerbation for at least three weeks
* Be stable
* Volunteering to participate in research
* To cooperate
* Patients with written consent form
* Healthy individuals in a similar age range without a diagnosed disease and symptoms will be included

Exclusion Criteria:

* Those with a history of chronic obstructive pulmonary disease exacerbations
* Individuals with orthopedic disease
* Individuals with neurological disease
* Individuals with other co-existing lung and systemic diseases other than chronic obstructive pulmonary disease
* Those who have had major surgery in the past few months
* Individuals with a history of recurrent significant clinical infections
* Have cognitive problems
* Having had unstable angina,
* Previous Myocardial Infarction
* Individuals with severe congestive heart failure refractory to medical therapy, individuals with uncontrolled hypertension
* Individuals with cancer

Ages: 40 Years to 75 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Chronic obstructive pulmonary disease (COPD) is a common, preventable and treatable disease characterized by persistent respiratory symptoms and airway limitation due to airway and/or alveolar abnormality resulting from exposure to harmful gases or particles and many factors that cause abnormal lung development.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Estimated)
Dates: Start 2021-07-20 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-05-20 (Estimated)

PRIMARY OUTCOMES:
Surface Electromyography | 45 minutes
  Activation of respiratory muscles will be performed with a surface Electromyography (EMG) device. The measurement will be performed by placing Electromyography (EMG) electrodes on the motor points of the respiratory muscles. Increased respiratory muscle activations indicate that respiratory muscles are used more; The decrease in respiratory muscle activations indicates that the respiratory muscles are used less.

SECONDARY OUTCOMES:
Measurement of Maximal Inspiratory Pressure | 5 minutes
  Maximal Inspiratory Pressure will be measured with an intraoral pressure measuring device. Maximal Inspiratory Pressure reflects respiratory muscle strength. An increase in Maximal Inspiratory Pressure indicates high respiratory muscle strength; A low Maximal Inspiratory Pressure value indicates respiratory muscle weakness.
Pulmonary Function Test | 5 minutes
  Pulmonary function test will be performed with a spirometer according to the criteria of the American Thoracic Society and the European Respiratory Society. While the decrease in pulmonary function test parameters shows worsening of lung functions; parameters in the normal range indicate good lung functions.
Chronic Obstructive Pulmonary Disease Assessment Test | 5 minutes
  Chronic Obstructive Pulmonary Disease Assessment Test is an eight-item scale measuring health status in Chronic Obstructive Pulmonary Disease. This scale is used to determine the health status of individuals with Chronic Obstructive Pulmonary Disease all over the world. Each question is scored between 0-5 and a total score between 0 and 40 is given. A score of 0 represents the best and a score of 40 represents the worst state of health.
Modified Medical Research Council Dyspnea Scale | 2 minutes
  It is a 5-item scale scored between 0-4 for individuals' shortness of breath. Evaluates dyspnea and activity limitation in individuals with chronic obstructive pulmonary disease. An increase in the score indicates an increase in shortness of breath.

CONTACTS AND LOCATIONS:
Locations (1):
- Bolu Abant İzzet Baysal University Department of Physiotherapy and Rehabilitation, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No